CLINICAL TRIAL: NCT06881641
Title: Sensitivity, Specificity, and Acceptability of a Bedside Formate Assay as a Diagnostic Tool in Methanol Poisoning: Prospective Observational and Randomized Studies
Brief Title: A Study on Bedside Formate Assay as a Diagnostic Tool in Methanol Poisoning
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC23008; NIHR203140 (Other: NIHR RIGHT4)
Record Dates: First submitted 2024-11-20; First posted 2025-03-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-02

CONDITIONS: Metabolic Acidosis
Keywords: methanol toxicity
MeSH Terms: conditions — Acidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Methanol poisoning is a serious issue, particularly in low- and middle-income countries (LMICs), where outbreaks can devastate communities. Diagnosing methanol poisoning is challenging because its symptoms mimic many other conditions, and traditional diagnostic methods require expensive lab equipment. Unfortunately, this often means doctors do not even consider methanol poisoning as a diagnosis. Methanol itself isn't highly toxic, but when the body breaks it down into formate, it becomes dangerous, leading to brain swelling and even death.

To address this, a study team has developed a new method to diagnose methanol poisoning using a single drop of blood with a device that can be used at the bedside, eliminating the need for any lab equipment. This point-of-care (POC) test measures formate, which is only present in cases of methanol poisoning.

The project consists of two sequential studies. The first study aims to compare the effectiveness of the POC formate test against standard lab tests, which can take several hours. The findings from this study will inform the second study.

The second study is a feasibility cluster randomized controlled trial. In this trial, entire hospitals, rather than individual patients, are randomly assigned different approaches, similar to tossing a coin. The goal is to determine whether this trial design can be used in larger-scale research to evaluate clinical outcomes. Specifically, it will examine whether the POC formate test can accelerate accurate diagnosis, enabling prompt treatment and preventing deaths.

DETAILED DESCRIPTION:
This study group has developed a new method for diagnosing methanol poisoning using a single drop of blood with a point-of-care (POC) device, eliminating the need for laboratory equipment. The device measures formate, present only in cases of methanol poisoning.

The research comprises two studies. The initial observational study (Study 1a) will assess the sensitivity and specificity of the POC formate assay compared to the laboratory formate assay (the gold standard). If the sensitivity is greater than 0.80, a feasibility three-arm cluster randomized controlled trial (RCT) (Study 1b) will follow to determine the feasibility of recruiting hospitals to a cluster RCT of formate diagnostic approaches.

This design will be used in the second study to test the clinical- and cost-effectiveness of incorporating the formate POC assay into routine clinical use.

Primary Objectives:

Study 1a: Determine the sensitivity and specificity of the POC formate assay compared to the laboratory formate assay.

Study 1b: Assess the feasibility of recruiting hospitals for a cluster RCT of formate diagnostic approaches.

Secondary Objectives:

Study 1a: Evaluate the use of the POC formate assay to identify methanol poisoning across diverse healthcare systems.

Study 1b: Compare clinical and resource use when introducing the POC formate assay into routine clinical practice.

Primary Endpoints:

Study 1a: Sensitivity and specificity of the POC formate test for diagnosing methanol poisoning.

Study 1b: Number of hospitals successfully recruited to the study.

Secondary Endpoints for Study 1a:

Time from patient arrival at the emergency department to sample collection.

Time from sample collection to result display by the POC assay and the laboratory assay.

Delay between result displays by the POC and the laboratory assay.

Time from sample collection until the clinician is informed of the results.

Time to initiation of antidote treatment and stopping unnecessary therapy in patients without methanol poisoning.

Secondary Endpoints for Study 1b:

Time to stopping unnecessary therapy in patients without methanol poisoning.

Proportion of patients with management changes based on the laboratory formate assay.

Clinical outcomes such as deaths, intubations, and dialysis needs.

Cost comparison between the POC formate assay, the laboratory assay, and no assay.

The study will include patients suspected of methanol poisoning or unexplained metabolic acidosis at large referral hospitals in Bangladesh and India. The study aims to determine whether the POC formate test can speed up the initiation of appropriate treatment, reduce unnecessary treatment costs, and improve clinical outcomes.

Study Population:

Patients presenting with suspected methanol poisoning or unexplained metabolic acidosis.

Number of Participants:

Study 1a: 1,620 participants.

Study 1b: 4,500 participants.

Inclusion Criteria:

Patients with suspected methanol poisoning or metabolic acidosis of unknown cause, including children aged 16-17 (with assent), adults (with consent), and those with relatives who can provide consent.

Exclusion Criteria:

Individuals unwilling to provide assent or consent.

Unaccompanied unconscious patients or those without a relative to provide consent.

Previously recruited individuals.

These studies aim to raise awareness of the methanol poisoning crisis, improve early detection and treatment, and establish high-quality protocols for patient care. They also aim to encourage junior doctors to pursue academic careers and practice good clinical habits. Raising awareness will help warn the public about dangerous alcohol and prevent further poisonings.

ELIGIBILITY:
Inclusion Criteria:

• Patients presenting with suspected methanol poisoning or metabolic acidosis of unknown cause, including:

* Children aged 16-17 years, who are willing to provide assent.
* Parents/Guardians of children who are able and willing to provide consent.
* Adults (aged 18 years with no upper age limit) who are willing to provide informed consent.
* Participants who lack capacity to consent for themselves but who have a relative who is willing and able to provide informed consent on behalf of the participant.

Suspected methanol poisoning will be based on clinician judgement using the following typical indicators of possible methanol ingestion:

1. History of:

   * Intake of illegal/bootleg/spurious alcohol, and/or
   * Other patients admitted with confirmed/suspected methanol poisoning and/or
   * Time from intake to symptoms >6-12 h
2. Symptoms/clinical findings

   * Coma, and/or
   * Hyperventilation (respiratory rate [RR] >20/min) and/or dyspnea, and/or
   * Visual disturbances (blurred vision, blindness), and/or
   * Gastrointestinal symptoms (vomiting, abdominal pain), and/or
   * Chest pain, and/or
   * Severe/unusual 'hang-over': Feeling very sick the following day, and/or
   * Pseudopapillitis

Metabolic acidosis of unknown origin will be based on the following features:

* Metabolic acidosis of unknown origin = origin not identified. The acidosis is not of unknown origin if the metabolic acidosis can be explained by another cause eg. lactic acidosis (e.g. where base deficit [BD] = 15 mM [i.e., base excess (BE) = -15 mM] and lactate is 12-15mM).
* An initial ABG shall be drawn. If the BD is >15mM (BE<-15mM), the patient shall be included (as long as "unknown origin" - see above). If the patient has a BD between 5-15, the acidosis is only moderate, and there is time to do the "fluid trial" (see below). If the acidosis improves within 1-2 hours after the fluid trial, the acidosis is unlikely to be because of methanol and the patient should not be included. If the acidosis does not improve, the patient should be included.

Exclusion Criteria:

* • Children aged 16-17 years, who are unwilling to provide assent.

  * Parents/Guardians of children who are unable or unwilling to provide consent.
  * Adults (aged 18 years with no upper age limit) who are unwilling to provide informed consent.
  * Participants who lack capacity to consent for themselves and who do not have a relative who is willing and able to provide informed consent on behalf of the participant (i.e. unaccompanied unconscious patients and others)
  * Individuals previously recruited to the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include patients presenting to large referral hospitals in 2 countries (Bangladesh, India) with suspicion of methanol poisoning or unexplained metabolic acidosis.
Sampling Method: Probability Sample
Enrollment: 6120 (Estimated)
Dates: Start 2025-06-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary objective 1 | Day1
  To determine the sensitivity and specificity of the POC formate assay compared to the laboratory formate assay.
Primary objective 2 | Day1
  Evaluate the use of the POC formate assay for methanol poisoning. Compare clinical and resource use of using the POC formate assay by introducing the assay into routine clinical use.

SECONDARY OUTCOMES:
Secondary objective | Day1
  Time interval (in minutes) from the patient's arrival at the emergency department until the sample is drawn from the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Michael Eddleston, Study Chair — University of Edinburgh
Locations (6):
- Bangladesh (5):
  - SZMCH, Bogra, Bogura
  - Rahshahi medical college hospital, Rajshahi, Rajshahi Division
  - Chittagong Medical College Hospital, Chittagong
  - Dhaka Medical College Hospital, Dhaka
  - Mag Osmania Medical College Hospital Sylhet, Sylhet
- PGIEMR, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided